CLINICAL TRIAL: NCT01005277
Title: Genetic Polymorphisms in ALL Samples Submitted to Gene Array Analysis
Brief Title: Study of Biomarkers in DNA Samples From Patients With Acute Lymphoblastic Leukemia or Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ABTR02B1; NCI-2009-00325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000271322; COG-ABTR02B1; ABTR02B1; ABTR02B1 (Other: Childrens Oncology Group); ABTR02B1 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2017-10

CONDITIONS: Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Adult Acute Promyelocytic Leukemia With PML-RARA; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia; Childhood Acute Myeloid Leukemia in Remission; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Ancillary-Correlative (genetic polymorphisms): Previously collected DNA samples are analyzed for polymorphisms at a variety of loci. Gene expression and expression profiles are correlated with genotype and therapy outcomes.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research study is looking at biomarkers in DNA samples from patients with acute lymphoblastic leukemia or acute myeloid leukemia. Studying samples of DNA from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Collect DNA samples from patients with cytogenetically, well characterized, and uniformly treated acute lymphoblastic leukemia or acute myeloid leukemia for use in analysis of a wide range of host factors influencing etiology and outcome of the disease.

II. Identify host factors that can be determined at onset of treatment to predict outcome of chemotherapy, and thus modify the therapy administered.

OUTLINE:

Previously collected DNA samples are analyzed for polymorphisms at a variety of loci. Gene expression and expression profiles are correlated with genotype and therapy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* DNA samples available from patients meeting the following criteria:

  * Infants with acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML)
  * Patients with pre-B ALL, including responders vs non-responders in selected genotypes [hyperdiploid, hypodiploid, t(12;21), t(9;22), t(1;19), and t(4;11)] and responders and non-responders regardless of genotype
  * Pediatric patients with AML registered on POG-9421
  * Adult patients with ALL, including t(8.21), inv(16), t(15;17), complex cytogenetics, and secondary AML
  * Pediatric patients with relapsed ALL enrolled on COG-AALL01P2
  * Pediatric patients enrolled on COG-9900 and other CCG or POG trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2002-04-17 (Actual); Primary Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Differences in induction outcome, dichotomized into complete remission or no remission | Up to 8 years
  Assessed with Fisher's exact test.
Differences in induction outcome, dichotomized into complete remission or no remission | Up to 8 years
  Assessed with Pearson's chi square statistic test
Differences in overall survival | Up to 8 years
  Evaluated using the log rank statistic.
Disease-free survival (DFS) | Time from the end of induction to relapse or death, assessed up to 8 years
  Evaluated using the log rank statistic.
Relapse-free survival | Time from the end of induction to marrow relapse or death from progressive disease, censoring on deaths from other causes, assessed up to 8 years
  Evaluated using the logrank statistic.
Etiology of leukemia: Chi square test | Up to 8 years
  Chi square test will be used to determine the differences in distribution of genotypes between cases and controls.
Etiology of leukemia: Fisher's exact test | Up to 8 years
  Fisher's exact test will be used to determine the differences in distribution of genotypes between cases and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, Principal Investigator — Children's Oncology Group
Locations (1):
- Childrens Oncology Group, Philadelphia, Pennsylvania, United States